CLINICAL TRIAL: NCT02960958
Title: Metabolome Analysis in Patients With Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Hee Koh, MD, The Catholic University of Korea
Other Study IDs: CiRAD1
Record Dates: First submitted 2016-11-08; First posted 2016-11-10 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: RheumatoId Arthritis
Keywords: Rheumatoid arthritis; Metabolomics; urine
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate discriminant metabolites in urine from patients with rheumatoid arthritis (RA) from healthy individuals. Then we determine if the patient's metabolic fingerprint could predict the development or flare-up of RA.

DETAILED DESCRIPTION:
Compare metabolites between RA patients and healthy individuals.

1. Collection urine sample
2. Assessing urine metabolites by 1H NMR spectroscopy
3. Analyzing the relationships between metabolites and clinical variables

ELIGIBILITY:
Inclusion Criteria:

* All patients with rheumatoid arthritis meet 2010 American College of Rheumatology/European League against Rheumatism classification criteria.

Exclusion Criteria:

* Comorbid with other autoimmune diseases
* Confirmed with amyloidosis
* Chronic kidney disease (estimated GFR < 60 ml/min/1.73m2)
* Chronic liver disease
* Thyroid disease
* Pregnancy
* Solid tumor/hematologic malignancy within 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with rheumatoid arthritis and healthy individuals
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11-20 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Metabolic fingerprint of rheumatoid arthritis | 1 years
  Metabolomic analyses of urine from patients with rheumatoid arthritis, healthy controls and other autoimmune disease

SECONDARY OUTCOMES:
Correlations between specific metabolites and disease activity/severity of RA | 1 year
  Identified metabolites and their clinical significances

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Koh, MD, Principal Investigator — Seoul St.Mary's hospital, The Catholic university of Korea

IPD SHARING:
Plan to Share IPD: No